CLINICAL TRIAL: NCT02356484
Title: Predictive Value of Surgical Stress Markers for Postoperative Complications: a Prospective Study
Brief Title: Surgical Stress Markers for Postoperative Complications: a Prospective Study
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, Professor, University of Lausanne Hospitals
Other Study IDs: 471/14
Record Dates: First submitted 2015-02-01; First posted 2015-02-05 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Operative Procedures, Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Major abdominal surgery cohort: In this surgical cohort, 4 inflammatory markers were measured: albumin, procalcitonin, CRP and lactate levels

SUMMARY:
The aim of this study is to evaluate the predictive value of albumine, C-reactive protein (CRP), procalcitonin, and lactates in terms of surgical stress and postoperative complications. These biomarkers will be measured from the day before surgery until postoperative day four in patients undergoing major surgery. Major surgery was defined as esophagus, gastric, liver, pancreas, endocrine, retroperitoneal, or colorectal procedures including an organ resection for benign or malignant disease and lasting more than 2 hours.

DETAILED DESCRIPTION:
This prospective study was conducted at the Department for Visceral Surgery at the University Hospital of Lausanne Switzerland (CHUV) between February and December 2015 (NCT02356484). The study was approved by the Institutional Review Board (No. 367/15), and all patients provided written consent prior to surgery. Inclusion criteria were age >18 years, and elective major abdominal surgery-defined as an operative procedure with anticipated duration ≥2 hours.17 Perioperative care closely adhered to recently published enhanced recovery guidelines (http://erassociety.org.loopiadns.com/guidelines/list-of-guidelines). Standardised fluid administration was followed by advanced haemodynamic monitoring to avoid intraoperative fluid overload. According to the clinical care pathway, intravenous fluid was typically discontinued the morning after surgery.

Biological markers Serum levels of albumin, CRP, PCT and lactate (LCT) were perioperatively measured in a fasting state, Following standardised institutional guidelines. Blood samples were drawn the day before surgery, the day of surgery (4-6 hours after the end of the operation) and on the first, second and third postoperative day. As Baseline values tend to show large variations especially for albumin,4 10 we considered that a dynamic value (difference between two time-points) might be more informative than a snapshot value. Several values based on preoperative and postoperative concentrations were thus calculated for each marker (ie, Δ Max: maximal difference between the preoperative and postoperative values; Δ POD 0: difference of concentration on POD -1 and POD 0; Δ POD 1: difference of concentration on POD-1 and POD 1).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients undergoing esophagus, gastric, liver, pancreas, endocrine, retroperitoneal, or colorectal surgery
* Operation time more than 2 hours
* Operation including an organ resection for benign or malignant disease

Exclusion Criteria:

* Immunosuppressive therapy
* Cognitive impairment or language comprehension problems
* Absence of the consent form prior to first blood sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major surgery (esophagus, gastric, liver, pancreas, endocrine, retroperitoneal, or colorectal surgery)
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hübner, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University of Lausanne Hospital, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Labgaa I, Joliat GR, Kefleyesus A, Mantziari S, Schafer M, Demartines N, Hubner M. Is postoperative decrease of serum albumin an early predictor of complications after major abdominal surgery? A prospective cohort study in a European centre. BMJ Open. 2017 Apr 8;7(4):e013966. doi: 10.1136/bmjopen-2016-013966. PMID 28391235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 inclusions planned 155 patients screened 17 refusals study stopped after 138 inclusions due to long recruitment time
Pre-assignment Details: From the 155 patients initially eligible for the study, 17 refused to participate, thus 138 patients were included in the study
Groups:
- Major Abdominal Surgery Cohort: One-arm study including all patients undergoing "major abdominal surgery according to the provided definition.
Period: Overall Study
Arm/Group | Major Abdominal Surgery Cohort
Started | 138
Completed | 138
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Major Abdominal Surgery Cohort
Number analyzed (Participants) | 138
Age, Continuous [Median (Full Range); unit: years] | 64 [50 to 73]
Sex: Female, Male [Count of Participants; unit: Participants] — demographical data such as patient gender were recorded
  Participants
    Female | 66
    Male | 72
Region of Enrollment [Number; unit: participants]
  Switzerland | 138

OUTCOME MEASURES:

1. Primary Outcome: Predictive Value of Postoperative Albumin Decrease in Terms of Surgical Stress and Postoperative Complications
Description: Delta albumin (g/l) before (day -1) and immediately (day 1) after surgery as a predictor of postoperative complications (until 30 days post surgery)
Time Frame: Albumin preoperatively (day -1) and postoperatively (day 1) after surgery
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Major Abdominal Surgery Cohort: Albumin was measured preoperatively and in postoperative day 1 for all 138 study participants
Arm/Group | Major Abdominal Surgery Cohort
Number analyzed (Participants) | 138
g/L | 11.3 (5.6)

ADVERSE EVENTS:
Groups:
- Major Abdominal Surgery Cohort: Patients undergoing major abdominal surgery according to the provided definition
Arm/Group | Major Abdominal Surgery Cohort
All-Cause Mortality (participants affected / at risk) | 1/138
Serious Adverse Events (participants affected / at risk) | 1/138
Other Adverse Events (participants affected / at risk) | 0/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Major Abdominal Surgery Cohort (N=138)
Cardiorespiratory arrest (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes